CLINICAL TRIAL: NCT02122731
Title: Southern Danish Hypertension and Diabetes Study (SDHDS) With Amiloride
Brief Title: Amiloride for Resistant Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ib Abildgaard Jacobsen (Other)
Responsible Party: Sponsor-Investigator, Ib Abildgaard Jacobsen, Consultant Physician, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2009-017033
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus; Microalbuminuria
Keywords: antihypertensive therapy; amiloride; add-on; resistant hypertension; blood pressure control; type 2 diabetes mellitus,; microalbuminuria.
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amiloride (Experimental): This is a non-randomized and non-controlled study with only one treatment arm with amiloride.
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Amiloride — 5 mg(daily of amiloride was added to patients triple antihypertensive therapy and increased to 10 mg/daily if office blood pressure at 4 weeks was above 130/80 mmHg.

SUMMARY:
To evaluate the antihypertensive effect of amiloride added to triple antihypertensive therapy in patients with resistant hypertension (RH) and type 2 diabetes mellitus (T2DM)

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the antihypertensive effect of amiloride added to triple antihypertensive treatment in patients with resistant hypertension and type 2 diabetes mellitus in an open-labelled, non- controlled and non-randomized interventional study.

The secondary objectives were to evaluate the additional effects of amiloride on:

* Urinary albumin excretion
* Blood pressure control, how many patients reached blood pressure control when amiloride was added to previous triple antihypertensive treatment.
* Plasminogen and plasmin excretion (ENaC activity) in the micro-and macroalbuminuric patients in the cohort.
* Urokinase plasminogen activator (uPA) activity

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with resistant hypertension (average daytime BP >130and/or >80 mmHg by ambulatory monitoring in spite of treatment with 3 antihypertensive drugs including a diuretic and an angiotensin coverting enzyme inhibitor (AECi) or angiotensin recpetor blocker (ARBs) and a third optional, all in optimal dosages.
* type 2 diabetes
* prior participant in a randomized controlled trial with spironolactone, but after a wash-out periods of minimum two weeks (NCT01062763)

Exclusion Criteria:

* Office blood pressure (BP) >180/110 mmHg
* daytime average BP by ambulatory monitoring > 170/85 mmHg
* heart failure (NYHA III-IV) Cardiac arrythmia HbA1C > 10% severe dyslipidemia known or with signs of secondary hypertension estimated glomerular filtration rate (eGFR) <50ml/min per 1.73 m2 prior intolerance to spironolactone or amiloride fertility without oral contraception pregnancy lactation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
average daytime systolic and diastolic blood pressure | 8 weeks
  ambulatory blood pressure monitoring was performed at baseline and after 8 weeks intervention with amiloride

SECONDARY OUTCOMES:
Urinary albumin excretion | after 8 weeks
  Urine albumin was measured at baseline and after 8 weeks of amiloride treatment.
plasma potassium | after 4 and 8 weeks
  plasma potassium tend to increase during amiloride treatment
urinary urokinase plasminogen activator (uPA) activity | At baseline and after 8 weeks of amiloride treatment
  uPA exist in urine where it cleaves plasminogen to plasmin. uPA is possible secreted fra the tubulus cells
urine plasminogen and plasmin | at baseline and after 8 weeks of amiloride treatment
  U-plasminogen is filtered to urine in patients with microalbuminuria. In urine plasminogen is activated to plasmin by urokinase plasminogen activator.Plasmin activates the epithelial sodium channel.

CONTACTS AND LOCATIONS:
Overall Officials: Ib A Jacobsen, DMSc, Principal Investigator — Odense University Hospital
Locations (4):
- Denmark (4):
  - Sydvestjysk Hospital, Esbjerg, Esbjerg
  - Sygehus Lillebaelt., Fredericia
  - Steno Diabetes Center, Gentofte Municipality
  - Odense University Hospital, Department of Endocrinology, Odense

REFERENCES:
- [Background] Oxlund CS, Henriksen JE, Tarnow L, Schousboe K, Gram J, Jacobsen IA. Low dose spironolactone reduces blood pressure in patients with resistant hypertension and type 2 diabetes mellitus: a double blind randomized clinical trial. J Hypertens. 2013 Oct;31(10):2094-102. doi: 10.1097/HJH.0b013e3283638b1a. PMID 24107738